CLINICAL TRIAL: NCT02278562
Title: Nutrition, Inflammation and Insulin Resistance in End-Stage Renal Disease
Brief Title: Nutrition, Inflammation and Insulin Resistance in End Stage Renal Disease-Aim 2
Acronym: INSPIRED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEPH-011-11S
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: ESRD
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Interleukin 1 Receptor Antagonist Protein; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- anakinra (Active Comparator): 100 mg of Anakinra in syringes administered subcutaneously 3 times a week for 3 months and lactose (placebo) in capsules administered orally 1 capsule per day for 3 months
  Interventions: Drug: anakinra
- actos (Active Comparator): Normal saline (placebo) in syringes administered subcutaneously 3 times a week for 3 months and 30 mg of Actos in capsules administered orally 1 capsule per day for 3 months
  Interventions: Drug: actos
- placebo 1 and 2 (Placebo Comparator): Normal saline (placebo) in syringes administered subcutaneously 3 times a week for 3 months and lactose (placebo) in capsules administered orally 1 capsule per day for 3 months
  Interventions: Other: placebo

INTERVENTIONS:
Drug: anakinra — 100 mg in syringes; administered subcutaneously 3 times a week for 12 weeks (3 months)
  Arms: anakinra
Drug: actos — 30 mg capsules; administered orally 1 capsule per day for 12 weeks (3 months)
  Arms: actos
Other: placebo — placebo capsules and injection
  Arms: placebo 1 and 2

SUMMARY:
By 2030 an estimated 2 million people in the US will need dialysis or transplantation for advanced kidney failure. An even more disturbing statistic is that mortality in End Stage Renal Disease (ESRD) is six times higher than in the general Medicare population with adjustment for age, gender and ethnicity. Protein energy wasting is highly prevalent in these patients and is one of the most important determinants of their poor clinical outcome.

Despite its well-recognized occurrence, the etiology and the mechanisms leading to protein energy wasting observed in chronic hemodialysis patients cannot be attributed to any single factor. However, irrespective of the specific etiologic mechanisms, it appears that the common pathway for all the metabolic derangements is related to exaggerated protein degradation relative to protein synthesis (47).

Two well-recognized and presumably interrelated metabolic abnormalities, insulin resistance and chronic inflammation, may be the major determinants of protein catabolism in coronary heart disease (CHD) patients. There are no studies examining the effects of anti-inflammatory interventions and/or insulin sensitizers on protein homeostasis in CHD. Due to their established anti-inflammatory and other pleiotropic effects, Interleukin-1 receptor antagonist Anakinra and insulin sensitizer peroxisome proliferator-activated receptors (PPAR) agonist Actos represent two such promising interventions. By modulating inflammatory response and insulin signaling through two pharmacological interventions, the investigators will have the unique opportunity to clarify mechanisms contributing of these two particular metabolic derangements in the development of protein energy wasting observed in chronic hemodialysis patients.

The overall goal is to elucidate the mechanisms by which chronic inflammation and insulin resistance influence the development of protein energy wasting in hemodialysis patients.

Specific Aim: To test the hypothesis that inhibiting inflammatory response by administration of an Interleukin1receptor antagonist (Anakinra) or increasing insulin sensitivity by administration of a PPAR agonist (Actos) will improve net protein metabolism.

Hypothesis: The chronic inflammatory component of protein energy wasting (PEW) observed in hemodialysis patients is, at least in part, mediated by insulin resistance.

Interim analysis may be performed (no specific plan at this time).

ELIGIBILITY:
Inclusion Criteria:

* Patients on CHD undergoing three time a week therapy for more than 6 months;
* Age 21 years old;
* Acceptable dialysis adequacy (spKt/V > 1.2);
* A patent, well-functioning, arterio-venous dialysis access;
* Ability to give informed consent;
* Life expectancy greater than 6 months;
* BMI >=20 and <=45.

Exclusion Criteria:

* Pregnancy;
* Intolerance or allergy to the study medication (including the metabolic clamp studies);
* Severe, unstable, active inflammatory disease (active infection, active connective tissue disorder), active cancer or cancer history in the prior 5 years except skin cancer, AIDS-HIV, active or history of liver disease (including hepatitis B virus and hepatitis C virus);
* Hospitalization or infection within 1 month prior to the study;
* Patients receiving steroids and/or other immunosuppressive agents (Prednisone > 5 mg/day; excluding inhaled and topical steroids);
* Diabetes Mellitus on insulin therapy;
* Previous history of tuberculosis (TB) with or without documented adequate therapy;
* Patients with recent close exposure to an individual with active TB;
* Females using oral contraceptives;
* Patients with New York Heart Association (NYHA) Class III or IV heart failure;
* Patients with a history of angina, myocardial infarction, transient ischemic attacks, or strokes within the last 6 months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Talat A Ikizler, MD, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN
Locations (1):
- Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ertuglu LA, Deger SM, Alsouqi A, Hung A, Gamboa J, Mambungu C, Sha F, Siew E, Abumrad NN, Ikizler TA. A randomized controlled pilot trial of anakinra and pioglitazone for protein metabolism in patients on maintenance haemodialysis. J Cachexia Sarcopenia Muscle. 2024 Feb;15(1):401-411. doi: 10.1002/jcsm.13395. Epub 2024 Jan 4. PMID 38178557

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at the VA Nashville and the Vanderbilt University Medical Center between October 2014 and March 2017.
Pre-assignment Details: There is about a 2-week screening period between enrollment and assignment to a treatment group to access inclusion/exclusion criteria. Although 33 subjects were enrolled, only 24 subjects were assigned to a treatment group (6 subjects were screen failures and 3 subjects withdrew prior to being randomized).
Period: Overall Study
Arm/Group | Anakinra | Actos | Placebo 1 and 2
Started | 9 | 7 | 8
Completed | 9 | 7 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anakinra | Actos | Placebo 1 and 2 | Total
Number analyzed (Participants) | 9 | 7 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (17) | 46 (15) | 56 (12) | 49 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 2 | 7
  Male | 5 | 6 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 9 | 7 | 7 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 6 | 7 | 19
  White | 3 | 1 | 1 | 5
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 7 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Leucine Disposal Rate (LDR)
Description: LDR is a sensitive laboratory assessment of amino acid metabolism
Time Frame: baseline and 3 months
Population: The number of participants for analysis was based on those subjects who completed the 3-month study. The analysis was per protocol.
Measure: Median (Inter-Quartile Range); unit: mg/kg/min
Arm/Group | Anakinra | Actos | Placebo 1 and 2
Number analyzed (Participants) | 9 | 7 | 8
mg/kg/min | -0.011 [-0.014 to -0.001] | 0.005 [-0.026 to 0.015] | 0.001 [-0.008 to 0.008]
Statistical Analysis 1: Comparison: Anakinra vs Placebo 1 and 2; Prior data indicate that LDR is normally distributed with standard deviation ranging from 0.16 to 0.23 in hemodialysis and control patients, respectively. If the true difference in the experimental and control means is 0.21, we will be able to reject the null hypothesis that the population means of the experimental and control groups are equal with probability (power) 0.933. The Type I error probability associated with this test of this null hypothesis is 0.05; Test type: Superiority; p = 0.37, Wilcoxon Rank-Sum — 0.05 is the a priori threshold for statistical significance
Statistical Analysis 2: Comparison: Actos vs Placebo 1 and 2; Prior data indicate that LDR is normally distributed with standard deviation ranging from 0.16 to 0.23 in hemodialysis and control patients, respectively. If the true difference in the experimental and control means is 0.21, we will be able to reject the null hypothesis that the population means of the experimental and control groups are equal with probability (power) 0.933; Test type: Superiority; p = 0.955, Wilcoxon Rank-Sum — 0.05 is the a priori threshold for statistical significance

2. Secondary Outcome: Change in Whole-body Net Protein Balance
Description: Whole-body net protein balance is the difference between protein synthesis (anabolism) and protein breakdown (catabolism) in the whole body
Time Frame: baseline and 3 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/kg/min
Arm/Group | Anakinra | Actos | Placebo 1 and 2
Number analyzed (Participants) | 9 | 7 | 8
mg/kg/min | -0.184 [-0.311 to -0.011] | -0.215 [-0.519 to 0.266] | 0.018 [-0.200 to 0.123]

3. Secondary Outcome: Change in Skeletal Muscle Net Protein Balance
Description: Skeletal muscle net protein balance is the difference between protein synthesis (anabolism) and protein breakdown (catabolism) in the skeletal muscles.
Time Frame: baseline and 3 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: μg/100 ml/min
Arm/Group | Anakinra | Actos | Placebo 1 and 2
Number analyzed (Participants) | 9 | 7 | 8
μg/100 ml/min | -5.1 [-47.9 to 79.2] | 11.8 [-34.7 to 26.6] | 134.1 [1.8 to 342.5]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Anakinra | Actos | Placebo 1 and 2
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 5/9 | 1/7 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra (N=9) | Actos (N=7) | Placebo 1 and 2 (N=8)
injection site reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
syncope (General disorders) | 2 (2) | 0 (0) | 0 (0)
allergic reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
fluid overload (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
access related (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
right side weakness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-12-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT02278562/Prot_SAP_000.pdf
  • Informed Consent Form (2015-06-02): https://cdn.clinicaltrials.gov/large-docs/62/NCT02278562/ICF_001.pdf